CLINICAL TRIAL: NCT06175247
Title: Low-Glycemic (LGI) Diet in Pregnant People With Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Epilepsy Foundation (Other)
Responsible Party: Principal Investigator, Regan J. Lemley, MD, Instructor of Neurology, Division of Epilepsy, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P001868
Record Dates: First submitted 2023-10-27; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Epilepsy
Keywords: low glycemic index diet; pregnancy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Glycemic Index Diet Group (Experimental): A low glycemic index diet will be started with ongoing dietician support & food questionnaires until pregnancy completion.
  Interventions: Other: Low Glycemic Index Diet
- Standard Diet Group (No Intervention): A standard diet, as chosen by participants, will be followed with ongoing food questionnaires until pregnancy completion.

INTERVENTIONS:
Other: Low Glycemic Index Diet — A low glycemic diet will be initiated with dietician support and guidance.
  Arms: Low Glycemic Index Diet Group

SUMMARY:
The goal of this clinical trial is to learn about the low glycemic index diet in pregnant people with epilepsy. The main questions it aims to answer are:

* Is the low glycemic index tolerable in pregnant people with epilepsy?
* Does the low glycemic index alter seizure frequency in pregnant people with epilepsy?
* Does the low glycemic index alter the gut bacteria & associated metabolic pathways in pregnant people with epilepsy? Participants will start the low glycemic index diet during pregnancy and will provide stool and blood samples a maximum of 3 times during study duration. Researchers will compare pregnant people with epilepsy on the diet to pregnant people with epilepsy not on a structured diet plan to see if tolerability, seizure frequency, and gut bacteria composition & metabolites differ.

DETAILED DESCRIPTION:
People with epilepsy who are planning for pregnancy or are pregnant have concerns about anti-seizure medication (ASM) treatment, as some ASMs increase the risk of major congenital malformations and can negatively influence cognitive outcomes in developing offspring (Tomson et al., 2018, Meador et al., 2021). Non-pharmacologic epilepsy treatments, such as specialized diets like the low glycemic diet or the modified Atkins diet, are not well studied in pregnant people with epilepsy but have proven to be effective in reducing seizures in the non-pregnant population. Dietary influence on seizure control is likely multifactorial, and recent studies have shown that one mechanism of action is to cause changes in the gut microbiome and alter neuroactive downstream bacterial metabolites, such as gamma-aminobutyric acid (Olson et al., 2018).

The low glycemic index (LGI) diet is one of the most flexible dietary therapies for epilepsy, and it appears to be safe in pregnancy with positive health outcomes for both the mother and baby (Walsh et al., 2012). Unfortunately, little is known about the effectiveness and mechanism of the LGI diet in pregnant patients with epilepsy. Therefore, the investigators propose this study in which the LGI diet will be initiated in the first half of pregnancy and explore LGI diet tolerability, seizure frequency, and potential underlying mechanisms in the pregnant epilepsy population.

Investigators will invite pregnant people with epilepsy up to 20 weeks gestation in the Brigham & Women's Epilepsy-Obstetrical clinic to participate in this study. Participants will choose to go on the low glycemic index diet or continue their standard diet, will a goal of enrolling 21 participants in a 1:2 intervention to control group ratio. Participants in the intervention group will meet will a dietician to initiate the diet and have ongoing dietician support and appointments. All participants will fill out diet questionnaires and provide a maximum of 3 stool samples and 3 blood samples. Dietary intervention will end when pregnancies end, and stool and blood samples will be collected up to 3 months postpartum. The main outcomes will be diet tolerability, seizure frequency, gut bacteria composition, and metabolite alterations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of focal or generalized epilepsy as defined by the International League Against Epilepsy
* Pregnant up to 20 weeks gestational age

Exclusion Criteria:

* Functional neurologic disorder
* Primary gastrointestinal disease
* Antibiotic use in past 3 months
* Diabetes
* Seizure freedom

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is based on gestational potential.
Enrollment: 21 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability of the low glycemic index diet in pregnant people with epilepsy | During the diet intervention and immediately after the diet intervention
  Tolerability will be measured by the number of participants able to continue the diet in pregnancy with diet questionnaires + dietician follow up visits.

SECONDARY OUTCOMES:
Seizure Frequency | Baseline pre-intervention, during the intervention, and through 3 months post-partum.
  Seizure Frequency in the 9 months prior to pregnancy & pre-enrollment will be determined via chart review, and seizures during pregnancy will be prospectively recorded. Pre-pregnancy and during pregnancy seizure frequencies will be compared.
Gut Bacteria Composition | During the intervention until 3 months postpartum
  Stool samples will be collected during and after pregnancy (maximum 3 samples per participant) in participants in each study group (experimental group on the low glycemic index diet, control group on regular diet). Samples will be sequenced, metagenomic libraries will be constructed and Quantitative insights for microbial ecology 2 (QIIME2) will be used to examine the magnitude of group differences.
Metabolic pathway alterations | During the intervention until 3 months postpartum
  Stool and blood samples will be collected during and after pregnancy (maximum 3 samples), metabolites will be identified, and metabolic pathway reconstruction will be performed to identify changes between participants in the experimental and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No